CLINICAL TRIAL: NCT02513069
Title: Mobile Contingency Management for Smoking Cessation in Returning US Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00050835
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Smoking; Veterans
MeSH Terms: conditions — Smoking | interventions — Nicotine Chewing Gum; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Contingency Management (mCM) (Experimental): The mCM arm represents a proactive tele-health intervention that combines guideline based cognitive-behavioral smoking cessation telephone counseling, a tele-medicine clinic for access to nicotine replacement therapy (NRT), and intensive behavioral therapy administered via a smart phone (with carbon monoxide monitor) based application. NRT may include nicotine patches (21 mg, 14 mg, and or 7 mg) used daily for six weeks from the smoking quit date. Dosage will depend on participants' reported smoking patterns and carbon monoxide readings. NRT may also include a "rescue" method, i.e., either nicotine gum or nicotine lozenge. The participants' preferred NRT rescue method will be prescribed and used as needed to reduce smoking craving for six weeks from the smoking quit date.
  Interventions: Other: Nicotine gum; Behavioral: mobile contingency management; Behavioral: Telephone counseling; Other: Nicotine patch; Other: Nicotine lozenge; Other: Smart phone; Other: Carbon monoxide monitor
- Tele-Health for Smoking Ccessation (Active Comparator): TELE-HEALTH FOR SMOKING CESSATION is a proactive tele-health intervention that will provide controls for therapist, medication, time and attention effects. The tele-health intervention provides the same guideline based cognitive-behavioral smoking cessation telephone counseling, and tele-medicine clinic for access to NRT as in the mCM intervention. NRT may include nicotine patches (21 mg, 14 mg, and or 7 mg) used daily for six weeks from the smoking quit date. Dosage will depend on participants' reported smoking patterns and carbon monoxide readings. NRT may also include a "rescue" method, i.e., either nicotine gum or nicotine lozenge. The participants' preferred NRT rescue method will be prescribed and used as needed to reduce smoking craving for six weeks from the smoking quit date.
  Interventions: Other: Nicotine gum; Behavioral: Telephone counseling; Other: Nicotine patch; Other: Nicotine lozenge

INTERVENTIONS:
Other: Nicotine gum — Participants will be prescribed one form of nicotine replacement "rescue" treatment (i.e., gum, lozenge), and may choose nicotine gum as the preferred "rescue" treatment. Participants will be instructed to use the rescue method as needed during the post-quit phase of the study to reduce cigarette cravings.
  Other Names: nicotine polacrilex
Behavioral: mobile contingency management — Participants will be asked to provide video recordings of themselves taking carbon monoxide readings in order to confirm smoking abstinence. Participants are asked to upload these videos to the study's secured server, and are provided reinforcement for videos that suggest smoking abstinence.
  Other Names: mCM
  Arms: Mobile Contingency Management (mCM)
Behavioral: Telephone counseling — Participants receive five sessions of cognitive-behavioral telephone counseling, and a participant manual. The telephone counseling protocol included in this application is based on standard cognitive-behavioral therapy techniques shown to be efficacious for smoking cessation and is informed by behavioral treatment principles .
  Other Names: CBT for smoking cessation
Other: Nicotine patch — Participants will be prescribed nicotine patches to be used during the post-quit phase of the study.
  Other Names: Nicoderm
Other: Nicotine lozenge — Participants will be prescribed one form of nicotine replacement "rescue" treatment (i.e., gum, lozenge), and may choose nicotine lozenge as the preferred "rescue" treatment. Participants will be instructed to use the rescue method as needed during the post-quit phase of the study to reduce cigarette cravings.
Other: Smart phone — Participants in the experimental condition will be loaned a smart phone to use during the mobile contingency management intervention period. The phone will be used to record videos of carbon monoxide readings to determine smoking abstinence.
  Arms: Mobile Contingency Management (mCM)
Other: Carbon monoxide monitor — Participants in the experimental condition will be loaned a CO monitor to use during the mobile contingency management intervention period. The monitor will be used to determine carbon monoxide content in the breath as a measurement of smoking.
  Other Names: CO monitor
  Arms: Mobile Contingency Management (mCM)

SUMMARY:
The primary goal of the study is to evaluate the effectiveness of a combined tele-health and contingency management (CM) intervention that the investigators call mobile CM, or mCM, in promoting smoking abstinence in US Veterans. The mCM intervention will combine a mobile system to reward non-smoking, smoking cessation counseling, and smoking cessation medications. The primary aim is to evaluate how effective this intervention is in promoting smoking abstinence compared to telehealth interventions for smoking cessation.

DETAILED DESCRIPTION:
Despite recent efforts to expand reach of smoking cessation treatment options beyond clinic based care, smoking cessation treatment including the use of smoking cessation aids remain greatly underutilized. If cessation programs are to have significant impact (Impact = Reach X Efficacy) on changing health behavior at the population level, there is a fundamental need to develop new and innovative strategies to increase treatment intensity, access, and participation. The use of intensive behavioral therapies, such as contingency management (CM), have demonstrated efficacy for reducing smoking in difficult-to-treat populations, but have had limited reach given the need to verify abstinence multiple times daily via clinic based monitoring. The development of a mobile health (mHealth) platform to provide CM has made the use of intensive CM approaches portable and feasible. The primary goal of the current study is to evaluate the effectiveness of a proactive tele-health intervention that combines evidenced based treatment for smoking cessation with smartphone based, portable contingency management on smoking rates. The central hypothesis is that increasing the intensity of available tele-health smoking approaches through the addition of mobile CM will be an effective way to reduce smoking rates in Veterans returning from the Iraq/Afghanistan wars. Guided by strong preliminary data, this hypothesis will be tested in a comparative effectiveness trial with a two-group design in which 260 Veteran smokers will be randomized to receive either an "mCM" intervention which combines evidence-based cognitive-behavioral telephone counseling (TC), a tele-medicine clinic for access to nicotine replacement (NRT), and mCM administered through a smart phone or to a control condition that will provide controls for therapist, medication, time and attention effects. Specific aims are to evaluate (1) the impact of mCM on rates of abstinence from cigarettes as measured by bio-verified, self-reported prolonged abstinence at 3-month, 6-month, and 12 month post-randomization follow-up, (2) the relative cost-effectiveness of the mCM intervention in quality adjusted life years (QALY), and (3) potential treatment mediators including self-efficacy and treatment process mechanisms. The approach is innovative because it builds upon advances in mHealth technology and will be the first evaluation of smart phone based mobile CM in conjunction with other evidence-based smoking cessation treatment for OEF/OIF/OND Veterans. There is a surprising lack of research aimed at evaluating multi-component smoking cessation interventions that integrate CM with evidence-based cognitive-behavioral treatment and smoking cessation aids such as NRT. Cigarette smoking remains the most lethal substance use disorder in the United States and military veterans are at particular high risk for smoking related morbidity and mortality. The significance of identifying cost-effective approaches to decreasing tobacco use in the relatively young and at-risk cohort of returning Veterans could be tremendous as it will prevent significant morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Smoked at least 10 cigarettes on at least 15 of 30 days before screening
* Served during OEF/OIF/OND era
* Are willing to make a smoking cessation attempt
* Enrolled in the Durham VA for ongoing care
* English speaking

Exclusion Criteria:

* Use and unwillingness to stop use of other forms of nicotine such as cigars, pipes, or chewing tobacco
* Active diagnosis of a primary psychotic disorder per medical record
* Are currently imprisoned or in psychiatric hospitalization
* Severely impaired hearing or speech such that telephone counseling is not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2015-01; Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
smoking, self-report | 6 month follow-up (6 months post-quit attempt)
  Participants' self-report of smoking in the past seven days will be measured at 6-month follow-up study visit.

SECONDARY OUTCOMES:
saliva cotinine | 6 month follow-up (6 months post-quit attempt)
  For participants reporting smoking abstinence at 6-months post treatment follow-up, the investigators will bio-verify smoking abstinence by collecting saliva samples that will be used to determine salivary cotinine levels.
smoking, self-report | Approx. ten weeks after enrollment (i.e., eight weeks after smoking quit attempt)
  Participants' self-report of smoking in the past seven days will be measured at approximately eight weeks after the participant's initial smoking quit attempt.
saliva cotinine | Approx. ten weeks after enrollment (i.e., eight weeks after smoking quit attempt)
  For participants reporting smoking abstinence eight weeks after their smoking quit attempt, the investigators will bio-verify smoking abstinence by collecting saliva samples that will be used to determine salivary cotinine levels.
smoking, self-report | 3 month follow-up (3 months post-quit attempt)
  Participants' self-report of smoking in the past seven days will be measured at 3-month follow-up study visit.
saliva cotinine | 3 month follow-up (3 months post-quit attempt)
  For participants reporting smoking abstinence at the 3-month follow-up contact, the investigators will bio-verify smoking abstinence by collecting saliva samples that will be used to determine salivary cotinine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S Calhoun, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States